CLINICAL TRIAL: NCT07097662
Title: Evaluation of the Effectiveness of Oxygen Reserve Index Monitoring During Pre-oxygenation in Obese Patients
Acronym: ORi
Status: Completed | Type: Observational
Sponsor: Irem Caner (Other)
Responsible Party: Sponsor-Investigator, Irem Caner, Research Assistant, Kocaeli University
Organization: Kocaeli University (Other)
Other Study IDs: KocaeliUIC
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In obese patients, the risk of perioperative complications such as rapid desaturation, atelectasis, difficult mask ventilation, difficult intubation, and hypoxia is higher compared to the normal population. Therefore, preoxygenation is even more critical in the obese patient group. In clinical practice, ETO2 is used as a practical indicator to evaluate sufficient oxygenation during preoxygenation. The Oxygen Reserve Index (ORiⓇ) is a new oxygenation monitoring parameter that is continuously and non-invasively measured by a specialized pulse oximetry device (Masimo, Irvine, CA).The primary objective of the investigators was to observe the correlation between ORIⓇ monitoring and ETO₂ during preoxygenation in obese patients.The secondary objective of the investigators was to evaluate the correlation of ORIⓇ with SpO₂ and PaO₂ in this patient population.

DETAILED DESCRIPTION:
Obesity is a chronic, progressive, and recurrent disease characterized by abnormal fat accumulation that adversely affects health and increases morbidity and mortality.

According to World Health Organization (WHO) data, the prevalence of obesity among adults aged 18 years and older is reported to be 16%.

Obese patients have an increased risk of perioperative complications compared to the general population, including rapid desaturation, atelectasis, difficult mask ventilation, difficult intubation, and hypoxia.

Therefore, preoxygenation is particularly important in obese patient populations.

The goal of preoxygenation is to maximize the duration during which the patient can tolerate apnea, thereby providing the anesthesiologist with crucial time to secure the airway in cases of planned or unanticipated "cannot ventilate, cannot intubate" scenarios.

In clinical practice, end-tidal oxygen concentration (ETO₂) is frequently used as a practical indicator to evaluate the adequacy of preoxygenation.

However, achieving a tight-fitting face mask and obtaining accurate ETO₂ measurements can sometimes be challenging.

Thus, alternative monitoring parameters may be needed to evaluate the effectiveness of preoxygenation.

The Oxygen Reserve Index (ORIⓇ) is a novel, continuous, and non-invasive oxygenation monitoring parameter provided by a specialized pulse oximeter (Masimo, Irvine, CA).

While SpO₂ is useful in assessing hypoxia and normoxia, and PaO₂ can evaluate a wide range of oxygenation states, arterial blood gas (ABG) analysis is limited due to its intermittent and invasive nature.

ORIⓇ offers real-time visibility into moderate hyperoxic states (PaO₂ between 100-200 mmHg), which SpO₂ cannot detect.

Several studies have investigated the use of ORIⓇ monitoring to evaluate preoxygenation efficacy in various patient populations.

It has been reported in the literature that ORIⓇ may serve as an early warning indicator of hypoxia and help predict unwanted hyperoxic episodes.

The primary objective of the investigators was to observe the correlation between ORIⓇ monitoring and ETO₂ during preoxygenation in obese patients.The secondary objective of the investigators was to evaluate the correlation of ORIⓇ with SpO₂ and PaO₂ in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a body mass index (BMI) >35 kg/m² scheduled for elective surgery
* ASA (American Society of Anesthesiologists) physical status classification I-III
* Patients aged 18 years and older

Exclusion Criteria:

* Patients with ASA physical status classification IV-V,
* Psychiatric disorders
* Severe cardiac arrhythmias
* Patients with an ejection fraction below 30%
* Chronic obstructive pulmonary disease (COPD)
* Those receiving home oxygen therapy
* Patients requiring supraglottic airway devices, and emergency cases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between February 2024 and July 2024, 60 patients aged 18 to 75 years, with an ASA physical status classification of II-III, a body mass index (BMI) greater than 35 kg/m², and scheduled for elective surgery under general anesthesia, were included in our study after obtaining verbal and written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Effectiveness of Oxygen Reserve Index Monitoring During Pre-oxygenation in Obese Patients | During 5-minute preoxygenation
  Non-invasive ORiⓇ values and ETO₂ levels measured every minute during tidal volume breathing in the preoxygenation period will be analyzed for correlation.

SECONDARY OUTCOMES:
Correlation between ORiⓇ and arterial oxygen pressure (PaO₂) at multiple time points after intubation | 30, 60, 90, and 120 minutes after intubation
  ORiⓇ values will be compared with simultaneously obtained arterial blood gas measurements (PaO₂) at predefined time points to assess correlation.
Correlation between ORiⓇ and peripheral oxygen saturation (SpO₂) at multiple time points after intubation | 30, 60, 90, and 120 minutes after intubation
  ORiⓇ values will be compared with corresponding SpO₂ measurements from pulse oximetry to evaluate correlation.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Caner, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hirata N, Nishimura M, Chaki T, Yoshikawa Y, Yamakage M. Comparison between oxygen reserve index and end-tidal oxygen concentration for estimation of oxygenation during pre-oxygenation via a tight-fitted face mask: A prospective observational study. Eur J Anaesthesiol. 2021 Mar 1;38(3):313-315. doi: 10.1097/EJA.0000000000001358. No abstract available. PMID 33538433